CLINICAL TRIAL: NCT06032988
Title: The Effect of Probiotic Supplements on Metabolic Control of People With Type 2 Diabetes in Greece. A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Probiotic Supplements on Metabolic Control of People With Type 2 Diabetes Mellitus in Greece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konstantinos Makrilakis, MD (Other)
Collaborators: Uni-Pharma (Industry)
Responsible Party: Sponsor-Investigator, Konstantinos Makrilakis, MD, Professor of Internal Medicine, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB approval No 306/26.04.2021
Record Dates: First submitted 2023-08-27; First posted 2023-09-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus type 2; Probiotics; Gut microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The present study will be a single-center, randomized, double-blind, placebo-controlled trial of a 6-month duration involving persons with T2D. Participants will receive either a multi-strain probiotic supplement (in the form of a capsule) or a matching placebo capsule once a day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned (using a computer generator [www.randomization.com], which randomizes each subject to a single treatment using randomly permuted blocks) to receive probiotic or placebo treatment, blinded to participants, study investigators, and physicians caring for the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LactoLevure (Active Comparator): The probiotic capsule LactoLevure^R will be given once a day
  Interventions: Dietary Supplement: LactoLevure
- Placebo (Placebo Comparator): Placebo capsules will consist of identical to the LactoLevure^R capsules of powdered glucose polymer, and will be given once a day
  Interventions: Dietary Supplement: LactoLevure

INTERVENTIONS:
Dietary Supplement: LactoLevure — Participants will receive LactoLevure^R probiotic dietary supplement or matching placebo once a day.
  Other Names: Probiotic

SUMMARY:
The goal of this interventional clinical study is to examine if there will be a change in metabolic indices (glycemic and lipid parameters) among persons with type 2 diabetes (T2D) who will receive a probiotic dietary supplement capsule for 6 months compared to those not receiving such a treatment (they will receive a matching placebo capsule that does not contain active ingredients).

The main questions to answer are:

1. Will glycemic indices, i.e., glycated hemoglobin (HbA1c) and fasting blood glucose, be different in people taking the probiotic treatment, compared to those not taking it, after 6 months?
2. Will other metabolic indices, mostly blood lipid levels (total cholesterol, triglycerides, HDL- and LDL-cholesterol) and liver function tests, be different in people taking the probiotic treatment compared to those not taking it after 6 months?
3. Will adiposity measures (weight, waist circumference) be affected by probiotic treatment in the two groups? Studies in animals and humans, mostly of shorter duration (<12 weeks) so far, have shown a possible trend towards improvement with probiotic treatment in all these parameters, but longer-term studies are scarce, and in Greece, there is none. Since diabetes treatment is complex (usually involving many medications) and expensive, developing cost-effective functional healthcare products for regulating blood glucose more efficiently has been recognized as a beneficial alternative.

Participants will be adult individuals (>18 years old) with T2D, followed at the outpatient Diabetes Center of the Laiko General Hospital, National and Kapodistrian University of Athens Medical School, in Athens, Greece, who will be randomized to receive either a probiotic dietary supplement or a matching placebo capsule, once a day. They will be followed every 3 months (as is customary for diabetic patients). They will be monitored regarding their glycemic control (HbA1c and fasting blood glucose), lipid parameters, liver and renal function, and anthropometric changes (weight, waist circumference, and blood pressure). Furthermore, participants will be asked to give a stool sample at the study's beginning and end (6 months) for gut microbiota analysis. A questionnaire will also be administered at the last visit (6 months) asking about patients' tolerance and satisfaction with the treatment (frequency of constipation, diarrhea, bowel function, bloating, gas production, and abdominal pain).

DETAILED DESCRIPTION:
Eligible participants will be randomized using a computer generator (www.randomization.com), which randomizes each subject to a single treatment by using the method of randomly permuted blocks, to receive either a multi-strain probiotic supplement (in the form of a capsule [LactoLevure^R]) or a matching placebo capsule, once a day. The probiotic capsule contains the species: Lactobacillus Acidophilus, Lactobacillus plantarum, Bifidobacterium lactis, Saccharomyces boulardii (in the following quantities of colony-forming units [CFU]: Lactobacillus Acidophilus 1.75x10^9 CFU, Lactobacillus plantarum 0.5x10^9 CFU, Bifidobacterium lactis 1.75x10^9 CFU, Saccharomyces boulardii 1.5x10^9 CFU). The capsules (probiotics brand name LactoLevure^R and placebo) are prepared and donated to the study personnel by an unrestricted research grant from Uni-Pharma Greece, the producer of LactoLevure^R (Uni-Pharma Pharmaceutical Laboratories S.A., Kifisia, Greece), who will have no other interference with the planning, the conduction, or the analysis of the results of the study. The probiotic and placebo capsules will have an identical appearance and packaging. Neither the participants nor the investigators will be aware of the treatment assignments in this double-blinded study. Additionally, participants will be asked not to change their diet and exercise habits and to refrain from consuming yoghurt or other similar dietary supplements during the study. Care will be taken not to change the other pharmaceutical medicines during the study (participants who will have to initiate insulin treatment will be excluded from further follow-up and analysis in the study).

Sample size calculation will be based on previous similar studies considering 80% power at α = 0.05 to detect a difference in metabolic indices. All participants will be given verbal and written information about the study and will sign an informed consent form according to the recommendations of the Declaration of Helsinki.

Participants will be seen every 3 months in the outpatient Diabetes center of the Laiko General Hospital, National and Kapodistrian University of Athens Medical School, in Athens, Greece (as is customary for diabetic patients) and will be monitored regarding their glycemic control (HbA1c and fasting blood glucose), lipid parameters, liver and renal function, and anthropometric variables changes (weight and waist circumference, blood pressure). Furthermore, participants will be asked to give a stool sample at the study's beginning and end (6 months) for gut microbiota analysis. A questionnaire will also be administered at the last visit (6 months) asking about patients' tolerance and satisfaction with the treatment (frequency of constipation, diarrhea, bowel function, bloating, gas production, and abdominal pain).

ELIGIBILITY:
Inclusion Criteria:

* T2D diagnosis of >6 months' duration
* Age 18-90 years
* A body-mass index (BMI) >18.5 kg/m^2
* HbA1c level >6 percent (%)
* on stable antidiabetic medications (oral or injectable glucagon-like peptide 1 receptor agonists [GLP-1 RAs]) for 8 weeks before the screening

Exclusion Criteria:

* Type 1 or other type of diabetes
* Pregnancy or wishing to become pregnant during the study
* End-stage kidney failure on dialysis, presence of other diseases, including cancer or severe hepatic insufficiency (transaminases >3.5x above normal)
* The use of other probiotic products or antibiotics over the previous 6 months
* Participation in other clinical trials
* Insulin administration
* The presence of other medical conditions that in the opinion of the investigators could jeopardize compliance with the protocol (e.g., malabsorption syndrome or an inability to take orally administered medications)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Effects of probiotics supplementation on glycemic control (HbA1c) | 6 months
  To measure the difference of the change from baseline in mean HbA1c (percentage points) between the intervention (probiotic) group and placebo, after 6 months

SECONDARY OUTCOMES:
Effects of probiotics supplementation on fasting blood glucose (FBG) | 6 months
  To measure the difference of the change from baseline of mean fasting blood glucose (FBG, mg/dl) between the intervention (probiotic) group and placebo, after 6 months
Effects of probiotics supplementation on lipid parameters (Total cholesterol, Triglycerides, HDL-C, LDL-C) | 6 months
  To measure the difference of the change from baseline of mean blood lipid levels, i.e. total cholesterol (mg/dl), triglycerides (mg/dl), HDL-cholesterol (mg/dl), LDL-cholesterol (mg/dl) between the intervention (probiotic) group and placebo, after 6 months. Any of these blood lipid measurements changes will be reported as lipid effects of the intervention.
Effects of probiotics supplementation on liver function tests (AST, ALT, γGT, Alkaline Phosphatase) | 6 months
  To measure the changes from baseline of mean blood liver function tests, i.e. AST (U/L), ALT (U/L), γGT (U/L) and Alkaline Phosphatase (U/L) between the intervention (probiotic) group and placebo, after 6 months. Any of these liver function test measurements changes will be reported as liver effects of the intervention.
Effects of probiotics supplementation on adiposity measures (BMI, Waist circumference) | 6 months
  To measure the difference of changes from baseline in adiposity characterisitcs (mean body mass index [BMI, kg/m^2] and/or mean waist circumference [cm]) between the intervention (probiotic) and placebo group after 6 months. Either or both of these adiposity measures changes will be reported as adiposity effects of the intervention.
Effects of probiotics supplementation on changes in gut microbiota diversity (alpha- and beta-diversity) | 6 months
  To measure the changes from baseline in stool microbial DNA diversity analyzed through 16S rRNA sequencing between the intervention (probiotic) and placebo group after 6 months. Alpha-diversity will measure the within-group changes in the richness (number) or distribution (evenness) of the microbial sample (in the intervention and the placebo group), whereas beta-diversity will measure the between-groups difference.

CONTACTS AND LOCATIONS:
Overall Officials: KONSTANTINOS MAKRILAKIS, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Laiko General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Individual participants' data will be deposited anonymized in "Pergamos", the central Institutional Repository of the National and Kapodistrian University of Athens
Time Frame: Within six months of completion of the study
Access Criteria: Anyone who wishes to access the data
URL: https://pergamos.lib.uoa.gr/uoa/dl/frontend/en/index.html

REFERENCES:
- [Background] Bock PM, Telo GH, Ramalho R, Sbaraini M, Leivas G, Martins AF, Schaan BD. The effect of probiotics, prebiotics or synbiotics on metabolic outcomes in individuals with diabetes: a systematic review and meta-analysis. Diabetologia. 2021 Jan;64(1):26-41. doi: 10.1007/s00125-020-05295-1. Epub 2020 Oct 13. PMID 33047170
- [Background] Rittiphairoj T, Pongpirul K, Janchot K, Mueller NT, Li T. Probiotics Contribute to Glycemic Control in Patients with Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis. Adv Nutr. 2021 Jun 1;12(3):722-734. doi: 10.1093/advances/nmaa133. PMID 33126241
- [Background] Vallianou NG, Stratigou T, Tsagarakis S. Microbiome and diabetes: Where are we now? Diabetes Res Clin Pract. 2018 Dec;146:111-118. doi: 10.1016/j.diabres.2018.10.008. Epub 2018 Oct 18. PMID 30342053